CLINICAL TRIAL: NCT01060306
Title: Prospective Optical cohereNce Tomography Evaluation of neoINtimal Coverage of a biodegrAdable Polymer-based Drug-eluting Stent
Brief Title: Optical Coherence Tomography Evaluation of a Biodegradable Polymer-based Drug-eluting Stent
Acronym: PONTINA
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: Ospedale Santa Maria Goretti (Other)
Responsible Party: Principal Investigator, Gregory Sgueglia, MD, MD, PhD, Ospedale Santa Maria Goretti
Other Study IDs: SMG-005
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bare metal stent 1 month: Patients implanted with the bare metal stent Gazelle evaluated for neointimal coverage one month after implantation
- Biodegradable polymer stent 6 months: Patients implanted with the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) evaluated for neointimal coverage after full drug elution and polymer biodegradation (6 months)
- Biodegradable polymer stent 7 months: Patients implanted with the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) evaluated for neointimal coverage one month after full drug elution and polymer biodegradation (7 months)

SUMMARY:
PONTINA aims at assessing by optical coherence tomography the neointimal coverage of the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) after full drug elution and polymer biodegradation (6 months), at one month after this time-point (7 months) and, as a comparator, of its bare metal stent counterpart (Gazelle stent) at 1 month after implantation.

ELIGIBILITY:
Inclusion Criteria:

* age >50 years
* de novo lesion
* lesion length <24 mm
* reference vessel diameter 3 mm

Exclusion Criteria:

* low compliance to dual antiplatelet therapy
* life expectancy <1 year
* allergy to any drug or substance use prior, during or after percutaneous coronary intervention
* chronic renal insufficiency
* low left ventricle ejection fraction (<35%)
* recent acute myocardial infarction
* previous coronary intervention
* off-label indication to stenting
* participation in another investigation
* refusal to participate to the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unstable coronary artery disease undergoing percutaneous coronary intervention on the left anterior descending artery with a Biomatrix stent placement or on the left circumflex artery with a Gazelle stent placement
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01 (Estimated); Primary Completion 2010-08 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of neointimal coverage of the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) after full drug elution and polymer biodegradation | 6 months

SECONDARY OUTCOMES:
Assessment of neointimal coverage of the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) one month after full drug elution and polymer biodegradation | 7 months
Comparison of neointimal coverage of the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) one month after full drug elution and polymer biodegradation and of its bare metal stent counterpart (Gazelle) one month after implantation | 7 months
Comparison of the neointimal coverage of the biodegradable polymer-based Biolimus A9-eluting stent (Biomatrix stent) after full drug elution and polymer biodegradation (6 months) and at one month after this time-point (7 months) | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Emodinamica e Cardiologia Interventistica - Ospedale Santa Maria Goretti, Latina, Italy